CLINICAL TRIAL: NCT07012616
Title: Supraclavicular Brachial Plexus Block as Opioid Sparing Technique in Pediatrics Undergoing Arteriovenous Fistula Creation: A Randomized Controlled Trial
Brief Title: Supraclavicular Brachial Plexus Block as Opioid Sparing Technique in Pediatrics Undergoing Arteriovenous Fistula Creation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1208/5/25
Record Dates: First submitted 2025-05-31; First posted 2025-06-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Supraclavicular Brachial Plexus Block; Opioid Sparing; Pediatric; Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraclavicular brachial plexus block group (Experimental): Patients will receive an ultrasound-guided supraclavicular brachial plexus block.
  Interventions: Other: Supraclavicular brachial plexus block
- Control group (No Intervention): Patients will not receive supraclavicular brachial plexus block as a control group.

INTERVENTIONS:
Other: Supraclavicular brachial plexus block — Patients will receive an ultrasound-guided supraclavicular brachial plexus block.
  Arms: Supraclavicular brachial plexus block group

SUMMARY:
This study aims to evaluate the efficacy of supraclavicular brachial plexus block as an opioid-sparing technique in pediatric patients undergoing arteriovenous fistula creation.

DETAILED DESCRIPTION:
The global incidence of end-stage renal failure (ESRF) is increasing. The preferred procedure for patients with ESRF undergoing maintenance Haemodialysis (HD) is the placement of an arteriovenous fistula (AVF).

In patients with ESRF, brachial plexus block (BPB) is frequently employed to administer anesthesia for the establishment or modification of AVF. This technique offers pain relief, sympathetic blockade, ideal surgical conditions, and a sufficient duration of postoperative block, preventing arterial spasms and graft thrombosis

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I- III.
* Undergoing arteriovenous fistula creation under general anesthesia.

Exclusion Criteria:

* Allergy to local anesthetics.
* Infection at the site of block.
* Local infection.
* Coagulation disorder.
* Previously failed or revision of blocked arteriovenous fistula.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperatively

SECONDARY OUTCOMES:
Total opioid consumption | 24 hours postoperatively
  Rescue analgesia of 0.5 µg/kg fentanyl will be given if the Wong-Baker score is 4 more.
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to the first dose of fentanyl administrated) will be assessed.
Degree of pain | 24 hours postoperatively
  Degree of pain will be assessed using Wong-Baker score (0 to 10), 0= no hurt and 10= hurts worst. Wong-Baker score will be assessed at post-anesthesia care unit (PACU), 4, 6, 8, 12, 18 and 24 h postoperatively.
Patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as local anesthetic systemic toxicity (LAST), bradycardia, hypotension, PONV, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.